CLINICAL TRIAL: NCT04379583
Title: HairDx Analytical Validation Study
Status: Withdrawn | Type: Observational
Why Stopped: Study no longer required by sponsor
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FI-HairDX-001
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-05

CONDITIONS: Hair Loss; Hair Loss/Baldness; Female Pattern Baldness; Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva DNA sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects: Female subjects providing DNA saliva sample
  Interventions: Device: HairDx Sample Collection Kit

INTERVENTIONS:
Device: HairDx Sample Collection Kit — Saliva collection using FDA OTC cleared sample collection device

SUMMARY:
The HairDx Test reports genetic variants associated with the development of FPHL.

DETAILED DESCRIPTION:
The HairDx Test reports genetic variants associated with the development of FPHL. The variants are detected from a saliva sample collected at home. The HairDx Test report is designed to help individuals understand the meaning of their results and encourage a conversation with a healthcare professional. The information provided by the HairDx Test report is not intended to start, stop or change any course of treatment. The purpose of this study is to collect DNA samples from subjects. The DNA samples will be used for the analytical validation of the HairDx Test. The results of this study will not be shared with the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females over the age of 18
* Overall good health
* Able to give informed consent
* Willing to collect saliva sample

Exclusion Criteria:

* Xerostomia (dry mouth)
* Inability to provide informed consent in English
* Inability to follow instructions for saliva sample collection
* Non US resident

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Female over the age of 18
Study Population: Female subjects recruited from an online advertisement approved by the IRB
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-06 (Estimated); Study Completion 2021-12-06 (Estimated)

PRIMARY OUTCOMES:
Determination of the accuracy of the HairDx Test | Baseline
  Determination of the accuracy of the HairDx Test in comparison to bi-directional Sanger sequencing
Determination of the precision and reproducibility of HairDx Test | Baseline
  Determination of the precision and reproducibility of HairDx Test in accordance with the laboratory instructions for use documentation

CONTACTS AND LOCATIONS:
Overall Officials: John McCoy, PhD, Principal Investigator — Applied Biology, Inc.
Locations (1):
- Applied Biology, Inc., Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with FDA.

REFERENCES:
- [Background] Redler S, Birch P, Drichel D, Hofmann P, Dobson K, Bohmer AC, Becker J, Giehl KA, Tazi-Ahnini R, Kruse R, Wolff H, Miesel A, Fischer T, Bohm M, Nuwayhid R, Garcia Bartels N, Lutz G, Becker T, Blume-Peytavi U, Nothen MM, Messenger AG, Betz RC. The oestrogen receptor 2 (ESR2) gene in female-pattern hair loss: replication of association with rs10137185 in German patients. Br J Dermatol. 2014 Apr;170(4):982-5. doi: 10.1111/bjd.12756. No abstract available. PMID 24344880